CLINICAL TRIAL: NCT02341469
Title: Integrated eDiagnosis Assessment (IeDA) for Children Under Five Years Old: a Stepped-wedge Randomized Cluster Trial of a Quality Improvement of the Management of Children Illnesses in Burkina Faso at the Primary Health Care Level
Brief Title: A Trial of an Integrated E-diagnosis Assessment to Improve the Management of Childhood Illnesses in Burkina Faso
Acronym: IeDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Terre des hommes, Burkina Faso & Switzerland - SPONSOR (Unknown); Centre Muraz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ITCRZC78
Record Dates: First submitted 2014-08-27; First posted 2015-01-19 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-10

CONDITIONS: IMCI Guidelines; Childhood Illnesses
Keywords: Burkina Faso; cluster randomised; stepped-wedge; IMCI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-of-care (No Intervention)
- integrated ediagnostic approach (Experimental)
  Interventions: Other: integrated ediagnostic approach (IeDA)

INTERVENTIONS:
Other: integrated ediagnostic approach (IeDA) — IeDA is a package of several interventions with the objective of improving the quality of child health care in health centres to ultimately decrease child morbidity and mortality. The components of IedA are described as follows:
  * REC: the IMCI protocol translated into a computer-based tool that aims to guide nurses during consultations.
  * The training of nurses on IMCI and REC.
  * A quality assurance mechanism through which each district and health centre is encouraged to find appropriate solutions in response to their local needs.
  * A supervision system conducted implemented by district managers to provide support and guidance to health centres.
  * A health information system based on data collected through the REC and fed back to the district managers and Heads of health centres.
  Arms: integrated ediagnostic approach

SUMMARY:
In 2010, one in six children in Burkina Faso died before the age of five, mainly due to lack of access to quality health care services. Most of these deaths could have been avoided through cost-effective interventions. Ensuring that sick children receive adequate care in a country where 80% of the population lives in rural areas requires improved accessibility and high quality primary health care services. The Integrated Management of Childhood Illnesses strategy (IMCI) was developed by the World Health Organization (WHO) and the United Nations Children's Fund (UNICEF) in the 1990s and is an excellent way to improve the quality of country's child health services. However, in Burkina Faso IMCI suffers from a low level of adherence by health workers. According to a recent evaluation by the Ministry of Health (MoH), only 8.2% of children had benefited in 2012 from an consultation using IMCI guideline. Moreover, an analysis of children's records showed that only 15% of IMCI consultations were being correctly delivered and, for instance, only 34% of children with pneumonia who needed an antibiotic were prescribed the correct treatment. The obstacles to IMCI adoption in Burkina Faso are diverse and include inadequate training methods, shortage of material (papers, forms), lack of quality supervision by district executive teams, lack of integration between IMCI monitoring tools and the national health information system etc.

The Integrated eDiagnosis Approach (IeDA) aims to address the poor quality of child health services in Burkina Faso by increasing the level of adherence to IMCI guidelines. IeDA is an innovative strategy combining information and communication technologies (using the Registre Electronique des Consultations [REC], an electronic IMCI patient record designed by Terre des hommes, Tdh) and a quality improvement approach. The approach has been piloted over three years in two different districts in the north of Burkina Faso, Tougan and Séguénéga. This medium scaling-up demonstration project will combine implementation and research components with a goal to enable national scaleup.

Terre des hommes is in charge of the implementation of the project and the London School of Hygiene and Tropical Medicine (LSHTM) will coordinate the research component of the study in partnership with Centre Muraz.

The primary hypothesis is that the Integrated eDiagnosis Approach will lead to improved adherence to IMCI guidelines and management of childhood illnesses in two regions (with a target of 75% of correct diagnoses and prescriptions).

ELIGIBILITY:
Inclusion Criteria:

Regions and Districts - The two regions Boucle du Mouhoune and Region du Nord were purposively chosen based on discussions with the MoH. Eight districts in these two regions will be included in the trial.

Health centres - Ten health centres in each district will be randomly selected and stratified so that, in each district, five health centres with fewer children aged 0-59 months than the district median and five health centres with more than the district median will be selected. The stratification reflects the variation in size between large and small health centres.

Patients - Children aged under five years old who attend the health centre for consultation at the day of the visit of the researchers.

Exclusion Criteria:

Health centres - All health centres not selected in the study will be excluded from the evaluation of the trial, but will still receive the intervention.

Patients - All children not present during the day of the visit of the researchers will be excluded. All patients above five years old will be excluded.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7200 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Adherence to IMCI guidelines | Three years
  Clinical observations will be conducted for children presenting at primary healthcare centres to determine the level of adherence to IMCI guidelines. This will be done at each step of the stepped-wedge trial, including at a baseline step (i.e. before any clusters are in the intervention phase).
Correct disease classification and prescription | Three years
  Following the clinical observation of each child, the child will be re-consulted by study staff to determine the correct disease classification(s) and prescription(s). A binary variable will be created for the consultation based on whether the classification(s) and prescription(s) decided by the healthcare worker are in agreement with those of our study staff.This will be done at each step of the stepped-wedge trial, including at a baseline step (i.e. before any clusters are in the intervention phase).

SECONDARY OUTCOMES:
Correct identification of danger signs | Three years
Correct classification of children | Three years
Prescription of the correct medicine | Three years
Correct referral or hospitalisation | Three years
Correct counselling delivered to child carer | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Karl Blanchet, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Centre Muraz, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Derived] Sarrassat S, Lewis JJ, Some AS, Somda S, Cousens S, Blanchet K. An Integrated eDiagnosis Approach (IeDA) versus standard IMCI for assessing and managing childhood illness in Burkina Faso: a stepped-wedge cluster randomised trial. BMC Health Serv Res. 2021 Apr 16;21(1):354. doi: 10.1186/s12913-021-06317-3. PMID 33863326
- [Derived] Blanchet K, Lewis JJ, Pozo-Martin F, Satouro A, Somda S, Ilboudo P, Sarrassat S, Cousens S. A mixed methods protocol to evaluate the effect and cost-effectiveness of an Integrated electronic Diagnosis Approach (IeDA) for the management of childhood illnesses at primary health facilities in Burkina Faso. Implement Sci. 2016 Aug 4;11(1):111. doi: 10.1186/s13012-016-0476-5. PMID 27488566